CLINICAL TRIAL: NCT00910676
Title: Phase II Multicentric Study About Preventive Treatment of Folliculitis Induced by the EGF-R Inhibitors in Patients With Metastatic Colorectal Cancer and Treated by Cetuximab or With Non-small-cell Lung Carcinoma Treated by Erlotinib
Brief Title: Study About Preventive Treatment of Folliculitis Induced by Epidermal Growth Factor Receptor Inhibitors
Acronym: DIPROCOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-002913-38; NCT00960388 (obsolete NCT alias)
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Colorectal Cancer; Non-Small-Cell Lung Carcinoma
Keywords: EGF-R inhibitors
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — betamethasone-17,21-dipropionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DIPROSONE (Experimental)
  Interventions: Drug: Diprosone

INTERVENTIONS:
Drug: Diprosone — * Start of treatment: as soon as the EGF-R inhibitors treatment begins
  * Application: On the body area susceptible to be affected by folliculitis, once a day, in the evening
  * Dosage: Quantity corresponded to around 2 tubes of 30 grams a week on the face, the chest and upper side of the back. There is no maximum dosage.
  * Period of treatment: 8 weeks

SUMMARY:
Patients will receive local prophylactic treatment (Diprosone cream) during 8 weeks from the beginning of the EGF-R inhibitors treatment, on the areas of the body susceptible to be affected by folliculitis.

ELIGIBILITY:
Inclusion Criteria:

* Indication of Cetuximab in patients with metastatic colorectal cancer in association or not with irinotecan, after failure of a chemotherapy treatment with Irinotecan OR
* Indication of Erlotinib, in patients with metastatic Non-Small-Cell Lung Carcinoma, after failure of at least one chemotherapy treatment
* No pre-existing cutaneous toxicity

Exclusion Criteria:

* Contraindication to local corticotherapy
* Previous history of severe hypersensibility reactions (Grade III or IV) due to Cetuximab, Irinotecan or Erlotinib
* Betamethasone or one of excipient product allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To reduce by 30 % the frequency of folliculitis by a local corticotherapy beginning at the same time that the treatment by EGF-R inhibitors began | 2 months of treatment by corticotherapy

SECONDARY OUTCOMES:
To assess the frequency of grade I, II and III folliculitis under Cetuximab and under Erlotinib | 2 months of treatment
To list the cutaneous side effects of the EGF-R inhibitors | 2 months of treatment
To assess the patient quality of life with the DLQI questionnaire | 2 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MORTIER, MD, Principal Investigator — Centre Hospitalier Régional et Universitaire de LILLE
Locations (3):
- France (3):
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Regional, Lille
  - Centre Hospitalier Régional, Lille